CLINICAL TRIAL: NCT05486598
Title: A Phase IB Clinical Trial to Evaluate the Effect of High-fat Diet on Pharmacokinetics of AL8326 Tablets in Chinese Healthy Adult Subjects
Brief Title: A Study of Diet Influence of AL8326 in Chinese Healthy Adult Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Advenchen Laboratories Nanjing Ltd. (Industry)
Responsible Party: Sponsor
Organization: Advenchen Laboratories, LLC (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AL8326-CN-009
Record Dates: First submitted 2022-06-02; First posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Diet, High-Fat; Pharmacokinetics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AL8326(Fasting） (Experimental): After screening, the subjects were randomly assigned to two sequence groups A and B. after fasting at least 10 hours overnight, they took al8326 tablets according to the requirements of two sequence groups A and B.
  Interventions: Drug: AL8326 tablets
- AL8326（Postprandial） (Experimental): After screening, the subjects were randomly assigned to two sequence groups A and B. after fasting at least 10 hours overnight, they took al8326 tablets according to the requirements of two sequence groups A and B.
  Interventions: Drug: AL8326 tablets

INTERVENTIONS:
Drug: AL8326 tablets — Sequence A group: on the 1st day, take a single dose of AL8326 tablets on an empty stomach. On the 15th day, take a single dose of AL8326 tablets after meals.
  Sequence B group: on the 1st day after meal, take a single dose of AL8326 tablets; on the 15th day, take a single dose of AL8326 tablets on an empty stomach.
  Other Names: AL8326

SUMMARY:
Main study objective: the pharmacokinetic effects of high-fat diet on AL8326 after oral administration of AL8326 tablets in Chinese healthy adult subjects.

Secondary study objectives: safety and tolerability of a single oral dose of AL8326 tablets in healthy subjects

DETAILED DESCRIPTION:
This is a Phase IB Clinical Trial to Evaluate the Effect of High-fat Diet on Pharmacokinetics of AL8326 Tablets in Chinese Healthy Adult Subjects.

Sixteen healthy subjects were randomly divided into two sequence groups, a and B, and eight subjects in each sequence group were dosed according to either the fasting → postprandial or the postprandial → fasting sequence. The washout period was 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects aged 18 ~ 65 years (including both 18 and 65 years);
2. Body weight ≥ 50 kg for men and ≥ 45 kg for women, with a body mass index in the range 19-26 kg / m^2 (inclusive 19 and 26) (BMI = body weight (kg) / height2 (M2));
3. No mental abnormalities, no history of cardiovascular, nervous, respiratory, digestive, urinary, endocrine and metabolic abnormalities;
4. Previous history, physical examination, vital signs, blood routine, urine routine, blood biochemistry, coagulation routine, pregnancy test (female), hepatitis, HIV, syphilis, 12 lead electrocardiogram, chest X-ray and other tests in the screening period, the whole of the results must be within the normal range matched to age and gender, or meet the protocol regulations, or if outside the normal range is judged as "not clinically significant (NCS) ";
5. Those who agree to be abstinent or have taken effective non drug contraception for the duration of the study and for at least 3 months after last study drug administration (for female subjects also required to be abstinent or have taken effective non drug contraception for two weeks prior to study entry);
6. Subject is able to communicate well with investigator and understand and comply with all requirements of this study, understand and sign the informed consent form.

Exclusion Criteria:

1. Allergic constitution (allergy to two or more substances) or known allergy to the study drug or to the same drug;
2. The screening period examination was abnormal and clinically significant.
3. Regular use of sedative, hypnotic, or other addictive drugs within 6 months before enrollment;
4. Those with a history of substance abuse or a positive urine drug abuse screen within 12 months prior to enrollment;
5. Those who smoked more than 5 cigarettes per day, or could not stop using any tobacco products during the trial;
6. Regular drinkers with a positive alcohol insufflation test or within 6 months prior to enrollment, who consumed more than 3 units of alcohol per day, or more than 21 units per week (one bottle of 350 ml of beer with 120 ml of liquor or 30 ml of spirits as 1 drinking unit);
7. Use of any prescription drug, Chinese herbal medicine within 4 weeks prior to enrollment, and / or use of any over-the-counter (OTC), food supplement (including vitamins, calcium tablets, etc.) within 2 weeks prior to first dose;
8. Had participated in other clinical trials and taken study drugs within 3 months before enrollment;
9. Having a blood donor (blood donation with ingredients) or blood loss of 400 ml, or having a blood transfusion within 3 months before enrollment; Blood donation (component containing blood donation) or blood loss of 200 ml within 1 month before enrollment (except physiological blood loss in females);
10. History of significant illness or major surgery, trauma, 3 months prior to screening.
11. Had gastrointestinal disease causing clinically significant symptoms such as nausea, vomiting, diarrhea, or malabsorption syndrome or a history of severe vomiting, diarrhea within the week prior to enrollment;
12. Pregnant, lactating female subjects and reproductive age female subjects unable to provide contraception on request;
13. Hepatitis B surface antigen positive, hepatitis C antibody positive, syphilis antibody positive, HIV antibody positive persons;
14. Special requirements for the diet (including lactose intolerance), inability to comply with the diet provided and respective prescribers;
15. Subject denied discontinuation of any beverage or food containing methylxanthine, e.g., caffeine (coffee, tea, cola, chocolate, etc.), 48 hours prior to first dose until the end of study;
16. Subject denied discontinuation of any beverage or food containing grapefruit 7 days prior to first dose until the end of the study;
17. Intolerance to venipuncture for blood collection or poor vascular status;
18. Subjects who, in the judgment of the investigator, were not suitable for participation in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
AUC0-t | 120 hours after each dose
  Effect of high fat diet on the pharmacokinetics of al8326 after oral administration of AL8326 tablets in Chinese healthy adult subjects.
AUC0-∞ | 120 hours after each dose
  Effect of high fat diet on the pharmacokinetics of al8326 after oral administration of AL8326 tablets in Chinese healthy adult subjects.
Cmax | 120 hours after each dose
  Effect of high fat diet on the pharmacokinetics of al8326 after oral administration of AL8326 tablets in Chinese healthy adult subjects.

SECONDARY OUTCOMES:
Tmax | 120 hours after each dose
  Safety and tolerability of a single oral dose of AL8326 tablets in healthy subjects.
T1/2 | 120 hours after each dose
  Safety and tolerability of a single oral dose of AL8326 tablets in healthy subjects.
Incidence of adverse events / serious adverse events as well as severity | Day 15 (± 1) after the last Administration
  Safety and tolerability of a single oral dose of AL8326 tablets in healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Cao, Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China